CLINICAL TRIAL: NCT02776488
Title: Exogenous Sodium Lactate Infusion in Traumatic Brain Injury (ELI-TBI)
Acronym: ELI-TBI
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The manufacturer of sodium lactate has stopped making the medication
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Paul Vespa, MD, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ELI TBI 1
Record Dates: First submitted 2016-05-13; First posted 2016-05-18 (Estimated); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Brain Injuries, Traumatic
Keywords: brain trauma, metabolic therapy
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Sodium Lactate; Saline Solution

STUDY DESIGN:
Intervention Model Description: Dose ranging and then RCT
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ELI Arm (Experimental): Infusion of exogenous sodium lactate as supplemental fuel within 48 hours of TBI
  Interventions: Drug: Sodium Lactate
- Placebo (Placebo Comparator): Placebo infusion of normal saline in Part 2 RCT
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium Lactate — Infusion of exogenous sodium lactate
  Arms: ELI Arm
Drug: Placebo — Infusion of normal saline
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
Metabolic crisis is a state of energy insufficiency due to impaired mitochondrial function as indicated by cerebral microdialysis lactate/pyruvate ratio (LPR). We have performed preliminary mechanistic analysis of alternative fuels in humans and have demonstrated proof of concept that exogenous fuels alter brain metabolism. We will conduct a multicenter, adaptive design-based, proof of concept phase 2 safety study of candidate supplemental fuels in patients with severe traumatic brain injury to determine safety and efficacy.

DETAILED DESCRIPTION:
Metabolic crisis is a state of energy insufficiency due to impaired mitochondrial function as indicated by cerebral microdialysis lactate/pyruvate ratio (LPR). We have performed safety analysis of exogenous sodium lactate infusions in humans and have demonstrated proof of concept that these fuels alter brain metabolism. Animal TBI studies have demonstrated proof of concept for exogenous lactate and pyruvate. We will conduct a multicenter, adaptive design-based, proof of concept biomarker mechanistic safety study of exogenous sodium lactate. The preliminary goal is to determine if exogenous lactate infusion is safe and has a demonstrated effect on selected biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients seen in the Medical Center Emergency Department
* Adult patients transferred to the Neurocritical Intensive Care Unit with a physician's diagnosis of brain injury.
* GCS 3-12

Exclusion Criteria:

* Pregnancy at time of injury
* History of diabetes mellitus
* History of hemodynamic instability
* Known terminal illness which alters brain functioning
* Diagnosed AIDS progressed to AIDS dementia
* Known history of chronic severe neurological disturbance
* Severe retardation
* Previous severe diminished mental capacity
* No command of either English or Spanish
* Arrest for a felony
* Active neurologic condition such as stroke, recent TBI
* metabolic disorder
* preexisting hyperlactatemia
* instability precluding experimental intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Mortality within 30 days | 30 days
  Percentage mortality within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Paul Vespa, MD, Principal Investigator — University of California Los Angeles, Department of Neurosurgery
Locations (1):
- David Geffen School of Medicine at UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
All protected health information (PHI) will be expunged from records before any sharing occurs

REFERENCES:
- [Background] Glenn TC, Martin NA, Horning MA, McArthur DL, Hovda DA, Vespa P, Brooks GA. Lactate: brain fuel in human traumatic brain injury: a comparison with normal healthy control subjects. J Neurotrauma. 2015 Jun 1;32(11):820-32. doi: 10.1089/neu.2014.3483. Epub 2015 Mar 31. PMID 25594628
- [Background] Glenn TC, Martin NA, McArthur DL, Hovda DA, Vespa P, Johnson ML, Horning MA, Brooks GA. Endogenous Nutritive Support after Traumatic Brain Injury: Peripheral Lactate Production for Glucose Supply via Gluconeogenesis. J Neurotrauma. 2015 Jun 1;32(11):811-9. doi: 10.1089/neu.2014.3482. Epub 2015 Mar 11. PMID 25279664
- [Background] Vespa P, McArthur DL, Stein N, Huang SC, Shao W, Filippou M, Etchepare M, Glenn T, Hovda DA. Tight glycemic control increases metabolic distress in traumatic brain injury: a randomized controlled within-subjects trial. Crit Care Med. 2012 Jun;40(6):1923-9. doi: 10.1097/CCM.0b013e31824e0fcc. PMID 22610193
- [Background] Vespa P, Bergsneider M, Hattori N, Wu HM, Huang SC, Martin NA, Glenn TC, McArthur DL, Hovda DA. Metabolic crisis without brain ischemia is common after traumatic brain injury: a combined microdialysis and positron emission tomography study. J Cereb Blood Flow Metab. 2005 Jun;25(6):763-74. doi: 10.1038/sj.jcbfm.9600073. PMID 15716852
- [Background] Vespa P, Tubi M, Claassen J, Buitrago-Blanco M, McArthur D, Velazquez AG, Tu B, Prins M, Nuwer M. Metabolic crisis occurs with seizures and periodic discharges after brain trauma. Ann Neurol. 2016 Apr;79(4):579-90. doi: 10.1002/ana.24606. Epub 2016 Feb 28. PMID 26814699
- [Background] Xu Y, McArthur DL, Alger JR, Etchepare M, Hovda DA, Glenn TC, Huang S, Dinov I, Vespa PM. Early nonischemic oxidative metabolic dysfunction leads to chronic brain atrophy in traumatic brain injury. J Cereb Blood Flow Metab. 2010 Apr;30(4):883-94. doi: 10.1038/jcbfm.2009.263. Epub 2009 Dec 23. PMID 20029449
- [Background] Bouzat P, Magistretti PJ, Oddo M. Hypertonic lactate and the injured brain: facts and the potential for positive clinical implications. Intensive Care Med. 2014 Jun;40(6):920-1. doi: 10.1007/s00134-014-3312-x. Epub 2014 May 1. No abstract available. PMID 24789621
- [Background] Bouzat P, Sala N, Suys T, Zerlauth JB, Marques-Vidal P, Feihl F, Bloch J, Messerer M, Levivier M, Meuli R, Magistretti PJ, Oddo M. Cerebral metabolic effects of exogenous lactate supplementation on the injured human brain. Intensive Care Med. 2014 Mar;40(3):412-21. doi: 10.1007/s00134-013-3203-6. Epub 2014 Jan 30. PMID 24477453
- [Derived] Vespa P, Wolahan S, Buitrago-Blanco M, Real C, Ruiz-Tejeda J, McArthur DL, Chiang JN, Agoston D, Glenn TC. Exogenous lactate infusion (ELI) in traumatic brain injury: higher dose is better? Crit Care. 2025 Apr 14;29(1):153. doi: 10.1186/s13054-025-05374-y. PMID 40229764